CLINICAL TRIAL: NCT06777212
Title: Mindfulness Intervention and Its Impact on Psychological and Family Dynamics in Children with Body-Focused Repetitive Behaviors.
Brief Title: Mindfulness Intervention for Psychological and Family Dynamics in Children with Body-Focused Repetitive Behaviors
Acronym: MIND-BFRB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ding Qiang, Intermediate Psychotherapist , Department of Fudan University Psychiatry and Psychology，Children's Hospital of FuDan University, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHFD-2025-01-BFRB
Record Dates: First submitted 2025-01-07; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Mindfulness Skills; Psychosocial Education
Keywords: Mindfulness Intervention; Body-Focused Repetitive Behaviors; Psychological Intervention; Nail-Biting; Skin-Picking; Hair-Pulling
MeSH Terms: conditions — Nail Biting; Excoriation Disorder; Trichotillomania

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: In this study, participants (children and their parents) will be unaware of the specific intervention group (Mindfulness Intervention or Psychosocial Education Control) they are assigned to after recruitment and consent. The random assignment to groups is managed entirely via the JingDong（JD） Health platform, and the interventions (daily mindfulness audio or psychosocial education articles) are delivered automatically through this platform. All outcome assessments (monthly and three-month follow-up surveys) will be conducted online via JD Health as well. Importantly, clinicians do not participate in the randomization, intervention delivery, or outcome assessments. Their role is limited to recruitment and initial consent collection. This ensures that clinicians are not involved in any part of the treatment or evaluation process, maintaining a fully masked design for participants and outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness intervention Group (Experimental): This group will receive a 30-day mindfulness intervention aimed at reducing Body-Focused Repetitive Behaviors (BFRBs) in children. The intervention includes daily mindfulness meditation exercises, such as deep breathing, body scans, and emotion awareness training, delivered via JD Health's platform. The children are encouraged to practice the exercises at home, with their parents providing support. The intervention is designed to improve emotional regulation, impulse control, and self-awareness in the participants. Assessments of behavioral and psychological outcomes will be collected at baseline, after one month, and at three months.
  Interventions: Behavioral: Mindfulness Training Program
- Psychosocial Education Control Group (Experimental): This group will receive a 30-day psychosocial education intervention aimed at improving emotional regulation and coping skills in children with Body-Focused Repetitive Behaviors (BFRBs). Daily educational content, including articles and coping strategies, will be delivered through JD Health's platform. Parents will assist in supporting and encouraging their children to engage with the educational materials. The program focuses on promoting family support, emotional awareness, and behavioral strategies. Behavioral and psychological assessments will be conducted at baseline, after one month, and at three months.
  Interventions: Behavioral: Psychosocial Education Program

INTERVENTIONS:
Behavioral: Mindfulness Training Program — The Mindfulness Training Program is a 30-day behavioral intervention designed to help children with body-focused repetitive behaviors (BFRBs) such as nail-biting, skin-picking, and hair-pulling. Delivered through JD Health, the program includes daily audio-guided exercises focused on mindfulness techniques such as deep breathing, body scans, and emotional awareness. Children will be encouraged to practice mindfulness for 10-15 minutes each day, with the goal of improving emotional regulation, reducing impulsive behavior, and enhancing self-awareness. Family support is involved, with parents helping children track their progress and offering reinforcement.
  Arms: Mindfulness intervention Group
Behavioral: Psychosocial Education Program — The Psychosocial Education Program is a 30-day behavioral intervention designed for children with body-focused repetitive behaviors (BFRBs), including nail-biting, skin-picking, and hair-pulling. Delivered through JD Health, the program provides daily educational content in the form of articles and coping strategies. The intervention focuses on improving emotional regulation, promoting family support, and developing positive behavioral strategies. Parents play an active role by reviewing the content with their children and helping them apply the strategies in daily life. Behavioral and psychological assessments are conducted at baseline, one month, and three months to evaluate the program's impact.
  Arms: Psychosocial Education Control Group

SUMMARY:
This is a single-center, randomized, controlled intervention study designed to evaluate the effectiveness of mindfulness intervention on reducing body-focused repetitive behaviors (BFRBs) in children aged 8-18, such as nail-biting, skin-picking, and hair-pulling. Participants will be randomly assigned to either a mindfulness intervention group or a psychosocial education control group. The study aims to assess the impact of the intervention on the severity and frequency of BFRBs, psychological health outcomes such as anxiety and depression, and family dynamics. Data will be collected through standardized psychological assessments. The study's findings will contribute to understanding the role of mindfulness in managing BFRBs and improving emotional and familial well-being in children.

DETAILED DESCRIPTION:
This study investigates the impact of mindfulness-based intervention (MBI) on children aged 8-18 with body-focused repetitive behaviors (BFRBs), including nail-biting, skin-picking, and hair-pulling. BFRBs often lead to psychological distress and impaired daily functioning. Current treatment options are limited, and mindfulness presents a promising non-invasive alternative. The study aims to evaluate the intervention's effectiveness in reducing BFRBs and improving psychological health and family dynamics. Participants will be randomized into two groups: a mindfulness intervention group and a psychosocial education control group. Both groups will participate in a 30-day program designed to address BFRBs, but with distinct approaches.

The mindfulness intervention group will engage in daily mindfulness exercises focusing on deep breathing, body scanning, emotional awareness, and behavior regulation for 10-15 minutes per day. The exercises are structured to build emotional awareness, manage impulses, and foster long-term emotional resilience. The program progresses through foundational mindfulness techniques, emotional acceptance, behavior modulation, and integrating mindfulness into daily life. Parents will actively participate by supervising and supporting their children's practice and recording their progress.

The psychosocial education control group will receive daily educational content designed to enhance emotional regulation and coping strategies. This content will be delivered via text and audio messages and will focus on improving emotional awareness, creating supportive home environments, and building healthy lifestyle habits. Parents will play a key role in implementing and supporting these strategies at home.

Baseline and follow-up assessments will be conducted to evaluate the intervention's effects on psychological health and family dynamics. Key measures include the frequency and severity of BFRBs as well as psychological health scales such as SCARED, CDI, OCI-CV ,s-EMBU-C and PHCSS. Parental mental health and family dynamics will also be assessed using validated tools, including the Conners Parent Rating Scale, SNAP-IV, PSI, and FAD. Assessments will be conducted at baseline (T0), immediately after the intervention (T1), and at a three-month follow-up (T2). Data analysis will focus on pre- and post-intervention comparisons to evaluate the mindfulness program's effectiveness in reducing BFRBs and improving emotional and family outcomes. Participants will be recruited from dermatology and psychiatric outpatient clinics at Children's Hospital of Fudan University . Recruitment will target children who have exhibited significant BFRBs within the last month, with informed consent obtained from their guardians.

ELIGIBILITY:
Inclusion Criteria:（1）Children and adolescents aged 8 to 18 years. （2）Evidence of significant Body-Focused Repetitive Behaviors (BFRBs) such as nail-biting, skin-picking, or hair-pulling, observed within the last month.

（3）Written informed consent provided by the parent or legal guardian, and child assent provided by the participant.

-

Exclusion Criteria:（1）Presence of severe physical illness or neurological disorders that may interfere with participation in the study.

（2）Participants currently receiving psychological interventions or pharmacological treatments for BFRBs or other psychiatric conditions, and who are unable to temporarily discontinue these treatments.

（3）Presence of significant cognitive impairment that would prevent the participant from completing study assessments or interventions.

-

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of Body-Focused Repetitive Behaviors (BFRBs) in Children as Reported by Parents | The primary outcome will be measured at baseline (pre-intervention), and at 1 month and 3 months after the intervention, based on parent assessments.
  The primary outcome measure will assess the severity of body-focused repetitive behaviors (BFRBs) in children, as reported by parents using the custom-designed BFRBS questionnaire. This questionnaire evaluates the frequency, duration, and distress caused by behaviors such as nail biting, skin picking, and hair pulling. The goal is to measure changes in the frequency and severity of these behaviors over the course of the intervention (Mindfulness Training or Psychosocial Education), with assessments at baseline, 1 month, and 3 months.
Severity of Body-Focused Repetitive Behaviors (BFRBs) in Children as Self-Reported by the Child | Baseline, 1 month, 3 months
  Children's self-reported experiences of BFRBs, including the frequency, duration, and distress, assessed through the custom-designed child version of the BFRBS questionnaire.

SECONDARY OUTCOMES:
Children's Depression Inventory (CDI) | Baseline (pre-intervention), 1 month post-intervention, 3 months post-intervention
  The CDI measures depressive symptoms in children, focusing on mood, behavior, and physical symptoms associated with depression. Scores range from 0 to 54, with higher scores indicating more severe depressive symptoms.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Baseline (pre-intervention), 1 month post-intervention, 3 months post-intervention
  The SCARED scale assesses the severity of anxiety symptoms in children, including subscales for separation anxiety, social phobia, generalized anxiety, panic, and specific fears. Scores range from 0 to 82, with higher scores indicating more severe anxiety symptoms.
Piers-Harris Children's Self-Concept Scale (PHCSS) | Baseline (pre-intervention), 1 month post-intervention, 3 months post-intervention
  The PHCSS measures children's self-concept, focusing on how they perceive themselves in domains such as behavior, emotions, and peer relationships. Scores range from 30 to 180, with higher scores indicating better self-concept and higher self-esteem.
Obsessive-Compulsive Inventory - Child Version (OCI-CV) | Baseline (pre-intervention), 1 month post-intervention, 3 months post-intervention
  The OCI-CV evaluates obsessive-compulsive behaviors in children, measuring both obsession and compulsion severity. Scores range from 0 to 36, with higher scores indicating more severe obsessive-compulsive behaviors.
Short Form of the Egna Minnen Beträffande Uppfostran(s-EMBU) | Baseline (pre-intervention), 1 month post-intervention, 3 months post-intervention
  The s-EMBU-C assesses children's perceptions of parental bonding and child-rearing practices, focusing on emotional support, rejection, and overprotection. Scores range from 1 to 5, with higher scores indicating better perceived parental bonding.
Parenting Stress Index (PSI) | Baseline (pre-intervention), 1 month post-intervention, 3 months post-intervention
  The Parenting Stress Index (PSI) assesses parental stress levels, focusing on areas such as child characteristics, parent characteristics, and the relationship between the parent and child.
  Scores range from 0 to 240, with higher scores indicating greater parental stress.
Conners Parent Rating Scale | Baseline (pre-intervention), 1 month post-intervention, 3 months post-intervention
  The Conners Parent Rating Scale is used to evaluate behaviors associated with Attention-Deficit/Hyperactivity Disorder (ADHD) in children. It includes a variety of behavioral and emotional issues that may indicate ADHD.
  Scores range from 0 to 60, with higher scores indicating more severe ADHD symptoms.
Swanson, Nolan, and Pelham Teacher and Parent Rating Scale - Version IV (SNAP-IV) | Baseline (pre-intervention), 1 month post-intervention, 3 months post-intervention
  The SNAP-IV scale measures attention and behavior issues, particularly related to ADHD. It is used to assess symptoms such as inattention, hyperactivity, and impulsivity, as observed by both parents and teachers.
  Scores range from 0 to 54, with higher scores indicating more severe attention and behavior issues.
The Family Assessment Device (FAD) | Baseline (pre-intervention), 1 month post-intervention, 3 months post-intervention
  FAD is a tool designed to assess family functioning, particularly focusing on communication and interaction patterns between family members. It evaluates various aspects of family life, such as communication, problem-solving, roles, affective involvement, behavior control, and general functioning. The FAD consists of 60 items, divided into several subscales that measure different aspects of family dynamics. The subscales include communication (the clarity and openness of communication between family members), problem-solving (the family's ability to resolve conflicts), roles (how responsibilities and roles are divided among family members), affective involvement (emotional support and connection between family members), behavioral control (discipline and structure), and general functioning (overall family cohesion and stability). Scores on the FAD range from 1 to 4, with higher scores indicating better family functioning and communication.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Ding, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared after publication of primary study results. Data will be de-identified to ensure participant confidentiality. Researchers can request access by submitting a proposal to the study team at [email address]. Approved researchers will receive access via a secure data-sharing platform.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date: 6 months after the publication of the primary study results. End Date: 5 years after the publication of the primary study results.
Access Criteria: Individual participant data and supporting information, including the study protocol, statistical analysis plan (SAP), informed consent form (ICF), clinical study report (CSR), and analytic code, will be made available to qualified researchers upon request. Access will be granted for academic and non-commercial purposes only.
  Researchers must submit a formal request to dingqiang@fudan.edu.cn, detailing their research objectives, study design, and ethical approval from an institutional review board (IRB) or ethics committee. Once approved, the requested data will be provided through secure channels, ensuring compliance with data privacy regulations and participant confidentiality. Access will be available for a period of 5 years following the publication of the primary study results.
URL: https://osf.io/dg5mf/files/osfstorage